CLINICAL TRIAL: NCT00851500
Title: A Trial of the Safety and Efficacy of K-604 for the Treatment of Atherosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Roger Morgan, MD Chief Medical Officer, Kowa Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-604-2.01US
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; carotid artery disease
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases | interventions — (2-(4-(2-benzimidazol-2ylthio)ethyl)piperazin-1yl)-N-(2,4-bis(methylthio)-6-methyl-3-pyridyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low dose K-604 (Experimental)
  Interventions: Drug: K-604
- high dose K-604 (Experimental)
  Interventions: Drug: K-604
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: K-604 — K-604 is given for 26 weeks
  Arms: high dose K-604; low dose K-604
Other: Placebo — placebo tablets are given for 26 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of K-604 for the treatment of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* moderate carotid artery stenosis

Exclusion Criteria:

* history of arteritis
* heavily calcified plaque
* uncontrolled hypertension
* poorly controlled diabetes
* hypercholesterolemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plaque composition over 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline in plaque size over 6 months. | 6 months

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Chandler, Arizona
  - Litchfield Park, Arizona
  - Phoenix, Arizona
  - Los Angeles, California
  - San Diego, California
  - Clearwater, Florida
  - Jacksonville, Florida
  - St Louis, Missouri
  - Buffalo, New York
  - Oklahoma City, Oklahoma
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Olympia, Washington
  - Renton, Washington
  - Seattle, Washington